CLINICAL TRIAL: NCT05072769
Title: The Effect of Date Consumption in the Early Postpartum Period on Uterine Involution
Brief Title: Date Consumption and Uterine Involution
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Dr. Kevser Ozdemir, PhD, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 48535046780
Record Dates: First submitted 2021-09-10; First posted 2021-10-11 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-09

CONDITIONS: Uterus Involution; Early Postpartum Hemorrhage
Keywords: birth; date fruit; oxytocin; uterus involution
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Chronology as Topic

STUDY DESIGN:
Intervention Model Description: There will be an experimental and a control group. Dates will be given to the experimental group after the birth, while the control group will be treated in line with the hospital routines.
Masking Description: There is no need for masking as placebo will not be applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): After the fetus and placenta are born, feeding 100 gr (5-6 pieces) dates to the experimental group
  Interventions: Dietary Supplement: Date Fruit
- Control group (No Intervention): The group that was not attempted any intervention in the postpartum period

INTERVENTIONS:
Dietary Supplement: Date Fruit — Within the first hour after birth, 100gr (5-6 pieces) dates will be eaten.
  Arms: Experimental group

SUMMARY:
There are many studies in the literature examining the effects of dates on pregnancy, birth and postpartum processes. However, no study has been found that examines the effect of women on the involution process in the early postpartum period. It is thought that this study will fill the gap in the literature with this study, which was conducted to determine the effect of date fed to women in the early postpartum period on uterine involution.

The study was planned as a randomized controlled and experimental study to determine the effect of date fed to women in the early postpartum period on uterine involution.

It will be held in the postpartum service of Sakarya University Training and Research Hospital between October - April 2021.

DETAILED DESCRIPTION:
There are many studies in the literature examining the effects of dates on pregnancy, birth and postpartum processes. However, no study has been found that examines the effect of women on the involution process in the early postpartum period. It is thought that this study will fill the gap in the literature with this study, which was conducted to determine the effect of date fed to women in the early postpartum period on uterine involution.

The study was planned as a randomized controlled and experimental study to determine the effect of date fed to women in the early postpartum period on uterine involution.

It will be held in Sakarya University Training and Research Hospital delivery room and postpartum service between October - December 2021.

The universe of the study will be women who gave vaginal birth between October and December 2021 in the delivery room and puerperal service department of Sakarya University Training and Research Hospital, and the sample will be 60 women (30 experimental group-30 control group).

Which of the women forming the sample group will be included in the experimental/intervention and control groups will be determined by simple randomization. A "random number generation program (research randomizer)" will be used in the randomization of the sample, and randomization with this program will be done by an unbiased researcher who is not involved in the research.

The implementation phase of the research will start after the third stage of labor (after the fetus and its appendages are born) ends. After the mother is stabilized, the "Descriptive Demographic Information Form" will be filled in for the experimental and control groups, and then blood samples will be taken from the mothers in order to determine the hemoglobin, hematocrit and oxytocin values. Since the blood sample will be taken from the intravenous line opened for emergencies during labor, an additional invasive procedure will not be applied to the patients. After the first blood sample is taken, 100gr (5-6 pieces) of Deglet Noor dates will be given to the experimental group and asked to be consumed within one hour. At this stage, the practices will continue in accordance with the hospital routines for the mothers in the control group. At the 6th hour after the third stage of labor, blood samples will be taken again to determine the hemoglobin, hematocrit and oxytocin values, and the application will end. In the postpartum ward, where the study will be conducted, routine blood samples are taken at the 6th hour after birth, so invasive intervention will be avoided.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the research,
* Primiparous,
* Not induction during birth,
* Born at term and healthy (38-42 weeks old, born 2500-4000gr, born with 5th minute apgar 7 and above, no known congenital disease),
* Not given oxytocin in the postpartum period,
* No oral intake restriction after controlling for postpartum uterine involution,
* Over 18 years of age who gave vaginal birth,
* It is planned to include mothers who can speak Turkish.

Exclusion Criteria:

* Not willing to participate in the research,
* Risk of postpartum bleeding in the first hour after delivery,
* Having a health problem in which the mother or baby is at risk,
* Not breastfeeding her baby
* Having a disease that prevents breastfeeding,
* Those whose hemoglobin value is below 10 g/dl,
* Cesarean delivery,
* Have a blood disease,
* The baby was taken to the neonatal intensive care unit,
* It is planned not to include mothers with diabetes.

Ages: 10 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin values | 6 hours
  Approximately 500 ml of blood is lost in vaginal delivery. Blood loss exceeding 500 ml in the postpartum period is a sign of bleeding. therefore, the involution process will be defined with the changes in hemoglobin (gr/dl) immediately after birth and 6 hours after birth.
Hematocrit values | 6 hours
  More than 10% decrease in the postpartum period compared to the prenatal period indicates bleeding. Therefore, the hematocrit (gr/dl) changes immediately after birth and 6 hours after birth will define the involution process.
Oxytocin values | 6 hours
  Oxytocin, which is produced in the hypothalamus and enters the circulation from the posterior pituitary, is a hormone that prevents postpartum hemorrhage by regulating the intensity and rhythm of postpartum uterine contractions. For this reason, the involution process will be defined by looking at oxytocin releases immediately after birth and 6 hours after birth.

CONTACTS AND LOCATIONS:
Overall Officials: Kevser Özdemir, Dr, Study Chair — Sakarya University
Locations (1):
- Sakarya University, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The study will be conducted with the data open to all researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be collected in the first hour and sixth hour after patients give birth. It will be reported after reaching the entire sample group.
Access Criteria: The data obtained from the study will be shared after it is reported and published.

REFERENCES:
- [Result] Razali N, Mohd Nahwari SH, Sulaiman S, Hassan J. Date fruit consumption at term: Effect on length of gestation, labour and delivery. J Obstet Gynaecol. 2017 Jul;37(5):595-600. doi: 10.1080/01443615.2017.1283304. Epub 2017 Mar 13. PMID 28286995
- [Result] Al-Kuran O, Al-Mehaisen L, Bawadi H, Beitawi S, Amarin Z. The effect of late pregnancy consumption of date fruit on labour and delivery. J Obstet Gynaecol. 2011;31(1):29-31. doi: 10.3109/01443615.2010.522267. PMID 21280989
- [Result] Kordi M, Meybodi FA, Tara F, Fakari FR, Nemati M, Shakeri M. Effect of Dates in Late Pregnancy on the Duration of Labor in Nulliparous Women. Iran J Nurs Midwifery Res. 2017 Sep-Oct;22(5):383-387. doi: 10.4103/ijnmr.IJNMR_213_15. PMID 29033994